CLINICAL TRIAL: NCT03942640
Title: Perineural Injection Therapy in Treatment of Chronic Supraspinatous Tendinopathy :A Randomized Clinical Trial Among Egyptian Patients .
Brief Title: Perineural Injection and Supraspinatus Tendenopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS.17.10.127
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-05

CONDITIONS: Supraspinatus Tendinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perineural injection group (Other): perineural injection therapy group (subcutaneous prolotherapy) This group included 30 patients aged from 18 to 60 years
  Buffered glucose preparation :
  2.4 ml of Na Bicarbonate 8.4% are mixed with 500ml dextrose 5%.
  Patients received 8 weekly injection sessions at sites of chronic constriction injurey of the following nerves :
  Suprascapular nerve..
  Interventions: Other: subctaneous perineural injection
- deepprolotherapy group (Other): Deep prolotherapy injection group The injection fluid contain 1 ml of 255 glucose and 1ml of lidocaine. The pathological area of the supraspinatous tendon was identified and graded using ultrasound pathology rating scale guided by ultrasonography (Simens Acuson p300 machine) Proper preparation with antiseptic solution of skin overlying the point of injection .
  Interventions: Other: deep prolotherapy

INTERVENTIONS:
Other: subctaneous perineural injection — Buffered glucose preparation :
  2.4 ml of Na Bicarbonate 8.4% are mixed with 500ml dextrose 5%. Patients received 8 weekly injection
  Arms: perineural injection group
Other: deep prolotherapy — The injection fluid contain 1 ml of 255 glucose and 1ml of lidocaine
  Arms: deepprolotherapy group

SUMMARY:
Atotal of 150 consecutive patients with chronic supraspinatous tendinopathy were invited to participate in the study .patients were recruited from the out patient clinic of rheumatology and rehabilitation department,Mansoura university hospital

a. perineural injection therapy group (subcutaneous prolotherapy) This group included 30 patients aged from 18 to 60 years Deep prolotherapy injection group The injection fluid contain 1 ml of 255 glucose and 1ml of lidocaine. The pathological area of the supraspinatous tendon was identified and graded using ultrasound pathology rating scale guided by ultrasonography (Simens Acuson p300 machine) Proper preparation with antiseptic solution of skin overlying the point of injection .

DETAILED DESCRIPTION:
Baseline Evaluation

All patients were subjected to the following:

1. Thorough History Taking

   1. Personal history: collected data include: age, sex, marital status, handedness, special habits and the current occupation.
   2. Complaint in the patient's own words.
   3. Present History he current symptoms, mode of onset, duration, , factors that may aggravate or relieve pain Characters of pain (dull aching,sharp pain ,burning sensation ,parasthesia). Distribution of pain . Review of systems: symptoms related to rheumatic conditions in particular conditions with predilection for shoulder joint affection.

      Symptoms suggestive of medical disorders e.g. diabetes mellitus or thyroid dysfunction.
   4. Past History Previous significant trauma(direct or occupational) orsugery to shoulder. Previous steroid injection to the shoulder. Previous injection of any type of regenerative medicine (as prp)
2. Thorough General Examination

   1. General condition.
   2. Vital signs (pulse, blood pressure, respiratory rate, body temperature)
   3. Examination of systems (chest,cardiovascular,abdominal,neurological) to identify medical condition that may cause shoulder pain.

      3-Muscloskeletal examination

   <!-- -->

   1. General muscloskeletal examination

Examination of all joints for :

I.deformity,visible swelling or muscle atrophy II.Palpation for tenderness,warmth,palpable swelling either bony enlargement or synovial effusion.

III.Abnormalities in range of motion. IV.Diffuse muscloskeletal pain. V.Abnormalities of gait.

ELIGIBILITY:
Inclusion Criteria:

Patients with supraspinatous tendinopathy

Exclusion Criteria:

-Shoulder joint instability omplete rotator cuff tear Adhesive capsulitis Septic arthritis Malignancy Coagulopathy Connective tissue diseases Spondyloarthropathies Previous corticosteroid injection in the last six months. Previous other forms of regenerative injection therapy (e.g prp injection therapy) in the last six mo

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
change of pain from baseline | immediately before injection,2 monthes after injection,3 monthes after injection
  The VAS-pain score is composed of a continuous horizontal line. This line is 100 mm in length. To measure the intensity of pain, the score is anchored by (0 score = no pain) at one end and (100 score = worst imaginable pain) on the other end. The patient places a mark to the VAS line at the point which represents the intensity of his pain
change of range of motion from base line | immediately before injection,2 monthes after injection,3 monthes after injection
  III.Examination of passive and active range of motion using goniometer based on the description of norkin and white as following
  * Abduction ;170
  * Adduction :50
  * Flexion :165
  * Extension:60
  * Internal rotation at 90 abduction :70
  * External rotation at 90 abduction :100

SECONDARY OUTCOMES:
change of function from base line | immediately before injection,2 monthes after injection,3 monthes after injection
  Shoulder pain and disability index : a self -administered questionnaire that consists of 2 dimentions ,one for pain and the other for functional activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Magdy Shaat, Al Mansurah, Dakahlia Provence, Egypt

IPD SHARING:
Plan to Share IPD: Undecided